CLINICAL TRIAL: NCT05457426
Title: Robotic Versus Laparoscopic Right Hemicolectomy With Complete Mesocolic Excision: a Retrospective Multicenter Study With Propensity Score Matching
Brief Title: Robotic Versus Laparoscopic Right Hemicolectomy With Complete Mesocolic Excision
Status: Completed | Type: Observational
Sponsor: Third Military Medical University (Other)
Responsible Party: Principal Investigator, Weidong Tong, Director of Gastrointestinal Surgery, Third Military Medical University
Other Study IDs: 20220623
Record Dates: First submitted 2022-06-23; First posted 2022-07-14 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Perioperative Outcomes; Oncological Outcomes
Keywords: Robot; Right hemicolectomy; Complete mesocolic excision

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- robotic right hemicolectomy with CME: The robot was set to come and dock from the right shoulder of the patient. Three robotic 8-mm trocars (R1, R2 and R3) and two 12-mm trocars (camera and assistant port) were used for the robotic procedure. One working arm carrying a monopolar cautery hook/scissors for dissection was located in the left upper quadrant port (R1). The other two working arms carried bipolar forceps in the suprapubic port (R2), and Cadiere's fenestrated forceps in the right lower quadrant port (R3) that was used to keep the superior mesenteric axis in traction. After gentle cephalad traction on the transverse mesocolon with the grasp in R3, the assistant grasped the ileocecal valve through the assistant port to put the ileocolic vascular pedicle on tension and the ileocolic vessels were identified and lifted up with R2. All procedures were performed keeping the principle of complete mesocolic excision.
  Interventions: Procedure: robotic right hemicolectomy with CME
- laparoscopic right hemicolectomy with CME: In the aparoscopic group, five trocars were used: a periumbilical incision and left upper quadrant for 12-mm trocars, both lower quadrants for 5-mm trocars, and the right quadrant for one more 5-mm trocar. A 30 degrees laparoscope was inserted through the periumbilical trocar site. After insertion of the trocars, the patient was placed in the Trendelenburg position with a 15 degrees rightward tilt. An ultrasonic device was used for dissection. All procedures were performed keeping the principle of complete mesocolic excision.

INTERVENTIONS:
Procedure: robotic right hemicolectomy with CME — The distribution of trocars was placed according to the position of Intuitive Surgical Inc. for robotic colectomy. The robot was set to come and dock from theright shoulder of the patient. Three robotic 8-mm trocars (R1, R2 and R3) and two 12-mm trocars (camera and assistant port) were used for the robotic procedure. One working arm carrying a monopolar cautery hook for dissection was located in the left upper quadrant port (R1). The other two working arms carried bipolar forceps in the suprapubic port (R3), and Cadiere's fenestrated forceps in the right lower quadrant port (R2) that was used to keep the superior mesenteric axis in traction. After gentle cephalad traction on the transversemesocolon with the grasp in R2, the assistant grasped the ileocecal valve through the assistant port to put the ileocolic vascular pedicle on tension and the ileocolic vessels were identified and lifted up with R3.
  Groups: robotic right hemicolectomy with CME

SUMMARY:
the investigators performed a retrospective multicenter propensity score matching study. From July 2016 to July 2021, 382 consecutive patients from different Chinese surgical departments were available for inclusion out of an initial cohort of 412, who underwent robotic or laparoscopic right hemicolectomy with CME.

DETAILED DESCRIPTION:
All consecutive patients who underwent robotic or laparoscopic right hemicolectomy with CME from July 2016 to July 2021 at three Chinese surgical departments (Department of General Surgery, Army Medical Center, Chongqing;Department of Colorectum, Chongqing University Three Gorges Hospital, Chongqing;Department of Colorectum, the 940th Hospital of Joint Logistics Support Force of Chinese People's Liberation Army, Lanzhou) were included in the study. A retrospective review of multicenter institutional database was conducted. The Da Vinci Surgical System (Intuitive Surgical, Sunnyvale, CA, USA) has been employed since 2016 in three centers. From July 2016 to July 2021, an initial cohort of 412 consecutive patients underwent robotic or laparoscopic right hemicolectomy with CME in three departments. With 30 cases meeting the exclusion criteria, 382 cases, including 204 males and 178 females, were available for inclusion. Of these, 149 cases by robotic right hemicolectomy with CME were classified as the robotic group, while the other 233 cases by laparoscopic right hemicolectomy with CME as the laparoscopic group.

ELIGIBILITY:
Inclusion Criteria:

1. Adenocarcinoma was confirmed by preoperative colonoscopy and it was located in the right colon.
2. Preoperative enhanced abdominal CT examination showed no invasion of abdominal wall or adjacent organs.
3. The patient underwent robotic or laparoscopic right hemicolectomy with CME.

Exclusion Criteria:

1. Multiple primary colorectal tumors
2. Metastasis to abdominal
3. Pelvic or distant organs
4. Accompanied with bowel obstruction or perforation
5. Neuroendocrine tumors
6. Lymphomas
7. Other malignant tumors.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients who underwent robotic or laparoscopic right hemicolectomy with CME from July 2016 to July 2021 at three Chinese surgical departments (Department of General Surgery, Army Medical Center, Chongqing; Department of Colorectum, Chongqing University Three Gorges Hospital, Chongqing; Department of Colorectum, the 940th Hospital of Joint Logistics Support Force of Chinese People's Liberation Army, Lanzhou) were included in the study
Sampling Method: Non-Probability Sample
Enrollment: 382 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-22 (Actual)

PRIMARY OUTCOMES:
diseasefree survival(months) | until July 2021
  Collect outcomes of follow-up and use Kaplan-Meier survival analysis to analyze it.
overall survival(months) | until July 2021
  Collect outcomes of follow-up and use Kaplan-Meier survival analysis to analyze it.

SECONDARY OUTCOMES:
conversion rates | during the surgery
  the incidence of a conversion to open surgery
operative time | during the surgery
  the miniutes of surgery from skin to skin
estimated blood loss | during the surgery
  the mililiter of the blood loss during surgery
oral retake | up to 30 days after surgery
  the patients begin to recover intake
time to return to bowel function | up to 30 days after surgery
  the patients begin to recover bowel function
length of stay | up to 30 days after surgery
  the days of hospital stay
total hospitalization cost | up to 30 days after surgery
  the total cost of this treatment by RMB
complications | up to 30 days after surgery
  Postoperative complications, such as ileus, anastomotic leak, small intestinal obstruction, bleeding and so on. Number of Participants with complications will be recorded.
harvest lymph nodes | up to 7 days after surgery
  the number of harvest lymph nodes in postoperative pathological report
lymph node metastasis | up to 7 days after surgery
  the number of patients with lymph node metastasis

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Chongqing University Three Gorges Hospital, Wanzhou, Chongqing Municipality
  - Army Medical Center, Yuzhong, Chongqing Municipality
  - No. 940 Hospital of Joint Logistics Support Foce of Chinese People's Liberation Army, Lanzhou, Gansu

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Yozgatli TK, Aytac E, Ozben V, Bayram O, Gurbuz B, Baca B, Balik E, Hamzaoglu I, Karahasanoglu T, Bugra D. Robotic Complete Mesocolic Excision Versus Conventional Laparoscopic Hemicolectomy for Right-Sided Colon Cancer. J Laparoendosc Adv Surg Tech A. 2019 May;29(5):671-676. doi: 10.1089/lap.2018.0348. Epub 2019 Feb 26. PMID 30807257
- [Result] Ferri V, Quijano Y, Nunez J, Caruso R, Duran H, Diaz E, Fabra I, Malave L, Isernia R, d'Ovidio A, Agresott R, Gomez P, Isojo R, Vicente E. Robotic-assisted right colectomy versus laparoscopic approach: case-matched study and cost-effectiveness analysis. J Robot Surg. 2021 Feb;15(1):115-123. doi: 10.1007/s11701-020-01084-5. Epub 2020 May 4. PMID 32367439
- [Result] Spinoglio G, Bianchi PP, Marano A, Priora F, Lenti LM, Ravazzoni F, Petz W, Borin S, Ribero D, Formisano G, Bertani E. Robotic Versus Laparoscopic Right Colectomy with Complete Mesocolic Excision for the Treatment of Colon Cancer: Perioperative Outcomes and 5-Year Survival in a Consecutive Series of 202 Patients. Ann Surg Oncol. 2018 Nov;25(12):3580-3586. doi: 10.1245/s10434-018-6752-7. Epub 2018 Sep 14. PMID 30218248